CLINICAL TRIAL: NCT00026923
Title: A Phase II Evaluation of Telesurgery Systems
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 990028; 99-C-0028
Record Dates: First submitted 2001-11-14; First posted 2001-11-15 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2001-12

CONDITIONS: Laparoscopy
Keywords: Laparoscopy; Telemedicine; Surgery; Endoscopy
MeSH Terms: interventions — Laparoscopy

INTERVENTIONS:
Procedure: Laparoscopic surgery

SUMMARY:
This study evaluates a system of remote supervision of laparoscopic surgery. Laparoscopic surgery is performed through small holes in the abdomen called ports. A camera is passed through one port for visualization. Laparoscopic surgery requires an assistant to hold the camera and help the operating surgeon view the surgical field. The assistant camera holder may be a surgeon or a robotic arm. The robotic arm is usually controlled by the operating surgeon. In this study, a robotic arm holding the camera will be used, and will be controlled by a surgeon outside the operating room.

DETAILED DESCRIPTION:
This study evaluates a system of remote supervision of laparoscopic surgery. Laparoscopic surgery is performed through small holes in the abdomen called ports. A camera is passed through one port for visualization. Laparoscopic surgery requires an assistant to hold the camera and help the operating surgeon view the surgical field. The assistant camera holder may be a surgeon or a robotic arm. The robotic arm is usually controlled by the operating surgeon. In this study, a robotic arm holding the camera will be used, and will be controlled by a surgeon outside the operating room.

ELIGIBILITY:
Any patient undergoing laparoscopic surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 1999-01; Study Completion 2001-12

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Kavoussi LR, Moore RG, Partin AW, Bender JS, Zenilman ME, Satava RM. Telerobotic assisted laparoscopic surgery: initial laboratory and clinical experience. Urology. 1994 Jul;44(1):15-9. doi: 10.1016/s0090-4295(94)80003-0. PMID 8042260
- [Background] Moore RG, Adams JB, Partin AW, Docimo SG, Kavoussi LR. Telementoring of laparoscopic procedures: initial clinical experience. Surg Endosc. 1996 Feb;10(2):107-10. doi: 10.1007/BF00188353. PMID 8932609
- [Background] Docimo SG, Moore RG, Adams J, Ben-Chaim J, Kavoussi LR. Early experience with telerobotic surgery in children. J Telemed Telecare. 1996;2 Suppl 1:48-50. doi: 10.1258/1357633961929259. No abstract available. PMID 9375090